CLINICAL TRIAL: NCT02739451
Title: A Randomised Controlled Trial of High-Flow Nasal Oxygen Versus Standard Oxygen Therapy in Critically Ill Immunocompromised Patients
Acronym: HIGH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM15003; P150912 (Other: Assistance Publique Hopitaux de Paris)
Record Dates: First submitted 2016-03-29; First posted 2016-04-15 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Acute Respiratory Failure
Keywords: immunocompromized patients; critically ill patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard oxygen group (Active Comparator): Oxygen therapy will be delivered using any device or combination of devices that are part of usual care: nasal oxygen, and mask with or without a reservoir bag and with or without the Venturi system
  Interventions: Procedure: standard oxygen
- High-flow nasal oxygen (HFNO) group (Experimental): Device that delivers humidified and warmed high-flow oxygen at flows greater than 15 L/min.
  HFNO will be initiated at a flow rate of 50 L/min and 100% FiO2. If the target SpO2 is not reached, the flow rate will be increased to 60 L/min. Then, FiO2 will be tapered to target an SpO2≥95. The minimal flow rate will be 45 L/min
  Interventions: Procedure: HFNO

INTERVENTIONS:
Procedure: standard oxygen — Devices used to treat spontaneously ventilating patients in the ICU who require supplemental oxygen. They deliver either
  * low-flow oxygen [including nasal cannula, Ventimask® without Venturi effect, and non-rebreather mask]
  * or medium-flow oxygen [Venturi masks and medium-flow facemasks]
  Arms: standard oxygen group
Procedure: HFNO — The intervention is the use of a device that allows to deliver high flow humidified and warmed oxygen. The device used is the Optiflow™ (Fisher&Paykel, Courtaboeuf, France).
  Arms: High-flow nasal oxygen (HFNO) group

SUMMARY:
Acute respiratory failure (ARF) is the leading reason for ICU admission in immunocompromised patients. Usual oxygen therapy involves administering low-to-medium oxygen flows through a nasal cannula or mask [with or without a bag and with or without the Venturi system] to achieve SpO2≥95%.

Oxygen therapy may be combined with non-invasive ventilation [NIV] providing both end-expiratory positive pressure and pressure support. However, in a recent trial by our group, non-invasive ventialtion [NIV] was not superior over oxygen without NIV.

High-flow nasal oxygen [HFNO] therapy is a focus of growing attention as an alternative to standard oxygen therapy. By providing warmed and humidified gas, HFNO allows the delivery of higher flow rates [of up to 60 L/min] via nasal cannula devices, with Fraction of inspired oxygen (FiO2) values of nearly 100%. Physiological benefits of HFNO consist of higher and constant FiO2 values, decreased work of breathing, nasopharyngeal washout leading to improved breathing-effort efficiency, and higher positive airway pressures associated with better lung recruitment.

Clinical consequences of these physiological benefits include alleviation of dyspnoea and discomfort, decreases in tachypnoea and signs of respiratory distress, a diminished need for intubation in patients with severe hypoxemia, and decreased mortality in unselected patients with acute hypoxemic respiratory failure However, although preliminary data establish the feasibility and safety of this technique, HFNO has never been properly evaluated in immunocompromised patients.

Thus, this project aims at demonstrating that HFNO is superior to low/medium-flow (standard) oxygen, minimising day-28 mortality

DETAILED DESCRIPTION:
After discussion at the investigator meeting and based on comments from the Data and Safety Monitoring Board on May 12, 2016, the DSMB has highlighted the need of the interim analysis (already planned) as benefits from high flow oxygen may be observed after 400 inclusions.

Update on June 16, 2017:

The number of patients enrolled is 488 and the inclusion rate is increasing steadily.

The interim analysis has been performed as scheduled and the DSMB decided that nothing should be changed.

ELIGIBILITY:
Inclusion Criteria:

* Known immunosuppression defined as one or more of the following: (a) immunosuppressive drug or long-term [>3 months] or high-dose [>0.5 mg/kg/day] steroids; (b) solid organ transplantation; (c) solid tumour; (d) haematological malignancy.
* ICU admission for any reason
* Need for oxygen therapy ≥6 Liters/min defined as one or more of the following: (a) respiratory distress with a respiratory rate >30/min; (b) cyanosis; (c) laboured breathing; (d) SpO2<90%; and (e) expected respiratory deterioration during a procedure
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Patient admitted to the ICU for end-of-life care. Do-not-intubate (DNI) patients can be included.
* Refusal of study participation or to pursue the study by the patient
* Hypercapnia with a formal indication for NIV [PaCO2 ≥ 50 mmHg, formal indication for NIV]
* Isolated cardiogenic pulmonary oedema [formal indication for NIV]. Patients with pulmonary oedema associated with another ARF etiology can be included.
* Pregnancy or breastfeeding
* Anatomical factors precluding the use of a nasal cannula
* Absence of coverage by the French statutory healthcare insurance system
* Post surgical setting from D1 to D6

After discussion at the investigator meeting and based on comments from the Data and Safety Monitoring Board on May 12, 2016, as all included patients need to have an acute hypoxemic respiratory failure and at least 6l of oxygen per minute, patients admitted to the ICU to secure any procedure (bronchoscopy etc..) or those not admitted for acute respiratory failure and who undergo intubation, will NOT be included in this trial. Only patients meeting criteria of acute respiratory failure will be included in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause day-28 mortality | 28 days

SECONDARY OUTCOMES:
Intubation or reintubation rate | days 3 and 28
  proportion of patients requiring invasive mechanical ventilation
patient comfort | 28 days
  Visual Analogue Scale (VAS) score
Intensity of dyspnoea | days 1-3
  Visual Analogue Scale (VAS) score
Perceived Exertion | days 1-3
  Borg scale
Respiratory rate | days 1-3
Oxygenation | days 1-3
  based on continuous saturation of peripheral oxygen (SpO2) monitoring, lowest SpO2 from D1 to D3 and PaO2/FiO2 on D1, D2, and D3
ICU length of stay | 28 days
Incidence of ICU-acquired infections | 28 days
Time to clear pulmonary infiltrates | 28 days
  Murray score
Oxygen-free and ventilation-free survivals | day 28
Re-intubation rate | day 28
Lowest median SpO2 during intubation | days 1-3
  for patients who were intubated during the study period
Repartition of acute mild/moderate/severe respiratory distress syndrome (ARDS) stages after intubation or reintubation as defined by the Berlin definition | day 28
Hypoxemic cardiac arrests | day 28
  After discussion at the investigator meeting and based on comments from the Data and Safety Monitoring Board on May 12, 2016, all hypoxemic cardiac arrests will be considered as suspected unexpected serious adverse reaction

CONTACTS AND LOCATIONS:
Overall Officials: Elie Azoulay, MDPhD, Principal Investigator — APHP
Locations (1):
- Medical ICU, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azoulay E, Lemiale V, Mokart D, Nseir S, Argaud L, Pene F, Kontar L, Bruneel F, Klouche K, Barbier F, Reignier J, Berrahil-Meksen L, Louis G, Constantin JM, Mayaux J, Wallet F, Kouatchet A, Peigne V, Theodose I, Perez P, Girault C, Jaber S, Oziel J, Nyunga M, Terzi N, Bouadma L, Lebert C, Lautrette A, Bige N, Raphalen JH, Papazian L, Darmon M, Chevret S, Demoule A. Effect of High-Flow Nasal Oxygen vs Standard Oxygen on 28-Day Mortality in Immunocompromised Patients With Acute Respiratory Failure: The HIGH Randomized Clinical Trial. JAMA. 2018 Nov 27;320(20):2099-2107. doi: 10.1001/jama.2018.14282. PMID 30357270
- [Derived] Azoulay E, Lemiale V, Mokart D, Nseir S, Argaud L, Pene F, Kontar L, Bruneel F, Klouche K, Barbier F, Reignier J, Stoclin A, Louis G, Constantin JM, Mayaux J, Wallet F, Kouatchet A, Peigne V, Perez P, Girault C, Jaber S, Oziel J, Nyunga M, Terzi N, Bouadma L, Lebert C, Lautrette A, Bige N, Raphalen JH, Papazian L, Rabbat A, Darmon M, Chevret S, Demoule A. High-flow nasal oxygen vs. standard oxygen therapy in immunocompromised patients with acute respiratory failure: study protocol for a randomized controlled trial. Trials. 2018 Mar 5;19(1):157. doi: 10.1186/s13063-018-2492-z. PMID 29506579